CLINICAL TRIAL: NCT03305172
Title: Structuring Financial Incentives to Increase Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Prof Ho Teck Hua, Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SG-STEP
Record Dates: First submitted 2017-09-26; First posted 2017-10-09 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity; Weight Loss
MeSH Terms: conditions — Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Subjects in the Control treatment are not given any financial incentive to achieve the goal.
- Gain Treatment (Experimental): Financial Incentive: Each subject in the Gain treatment will earn a certain amount of money for each day the goal is achieved. The money earned will be added to a virtual account that the subject has, and will be paid to the subject at the end of the intervention period.
  Interventions: Behavioral: Financial Incentive
- Loss Treatment (Experimental): Financial Incentive: Each subject in the Loss treatment will be given a certain amount of money in his/her virtual account at the beginning of every week. For each day that the subject does not achieve the goal, a small portion of that money will be deducted from the virtual account. The balance that is left in the virtual account will be paid to the subject at the end of the intervention period.
  Interventions: Behavioral: Financial Incentive
- Gain Streak Treatment (Experimental): Financial Incentive: Each subject in the Gain Streak treatment get an increasing amount of money added to his/her virtual account for every continuous day that they achieve the goal. The maximum cumulative amount per week is same as in the other treatment conditions. The payment is reset at the beginning of each week, or if the subject misses the goal on any day. The money in the virtual account will be paid to the subject at the end of the intervention period.
  Interventions: Behavioral: Financial Incentive
- Loss Streak Treatment (Experimental): Financial Incentive: Each subject in the Loss Streak treatment will be given a certain amount of money in his/her virtual account at the beginning of every week. An increasing amount of money will be deducted for each consecutive day the subject does not achieve the goal. The payment is reset at the beginning of each week, or when the subject achieves the goal (i.e., deductions are reset when the streak is broken). The balance that is left in the virtual account will be paid to the subject at the end of the intervention period.
  Interventions: Behavioral: Financial Incentive

INTERVENTIONS:
Behavioral: Financial Incentive — Giving different structures of long term (36 weeks) financial incentives to increase physical activity
  Arms: Gain Streak Treatment; Gain Treatment; Loss Streak Treatment; Loss Treatment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of different structures of long term financial incentives on increasing physical activity performed by subjects, as measured by the number of steps walked per day.

Investigators are interested in studying whether physical activity increases during an intervention period (with incentives) and a post-intervention period (with no incentives).

DETAILED DESCRIPTION:
The proposed study is a field experiment. Adults within the ages of 25 and 60 years of age, and with a body mass index of 22 or higher will be eligible to participate.

The study will consist of (1) a two-week baseline period, (2) a 36-week intervention period, and (3) a 12-week follow-up period.

At the beginning of the study, subjects will be given a wearable fitness device and their daily step count will be monitored for two weeks; this is the baseline period. After the two-week baseline period, the subjects will be randomly assigned to one of the five different conditions (Control, Gain, Loss, Gain Streak, or Loss Streak) and will be given the goal to increase their baseline step counts by 2,500 steps.

=====

HYPOTHESES -- Investigators expect the following:

1. Loss Aversion: Subjects in the Loss treatment will achieve the goal on a greater number of days than subjects in the Gain treatment.
2. Streak: Subjects in the Gain treatment will achieve the goal on a greater number of days than subjects in the Gain Streak treatment.
3. Loss Streak: Subjects in the Loss treatment will achieve the goal on a greater number of days than subjects in the Loss Streak treatment. Whether subjects in the Loss Streak treatment will perform better or worse than subjects in the other two treatments will be investigated.

CONTRIBUTION -- Prior research has not examined the effect of a long term financial incentive (36 weeks) on individual behavior in achieving a goal. In this study, the investigators also examine two additional financial incentive structures: Gain Streak and Loss Streak. If the hypotheses are correct, the results have important implications for designing financial incentives to encourage good behavior and to encourage good habit formation across domains.

ELIGIBILITY:
Inclusion Criteria:

* Singapore citizens and permanent residents
* Adults with BMI greater than 22
* Ownership of a smartphone or tablet
* Only one member per household can participate in the study

Exclusion Criteria:

* Women who are pregnant or breast feeding, or who intend to become pregnant over next year
* Subjects who are already participating in another physical activity program or study
* Subjects who are unable to participate for a total of 1 year
* Subjects who are unwilling to wear the fitness device
* Subjects who already walk more than 10,000 steps a day (self-reported per-day-average over seven days)
* Subjects who have any of the following health conditions:

  * high blood pressure
  * high cholesterol
  * heart attack
  * heart failure
  * stroke
  * chronic obstructive pulmonary disease
  * kidney disease
  * diabetes (type 2)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 620 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Step count goal -- Intervention | 36-week intervention period following the baseline period.
  Proportion of participant-days on which the goal (baseline +2,500 steps) was achieved during the intervention period.
Change in mean daily steps -- Intervention | 36-week intervention period following the baseline period.
  Change in mean daily steps during the intervention period.

SECONDARY OUTCOMES:
Step count goal -- Post-intervention | 12-week post-intervention period.
  Proportion of participant-days on which the goal (baseline +2,500 steps) was achieved during the post-intervention period.
Change in mean daily steps -- Post-intervention | 12-week post-intervention period.
  Change in mean daily steps during the post-intervention period.
Sleep Pattern -- Intervention | 36-week intervention period following the baseline period.
  Changes in sleep pattern (deep sleep, hours of continuous sleep) during the intervention period.
Sleep Pattern -- Post-intervention | 12-week post-intervention period.
  Changes in sleep pattern (deep sleep, hours of continuous sleep) during the post-intervention period.
Weight (in kilograms) Loss -- Intervention | 36-week intervention period following the baseline period.
  Drop in weight from baseline to the end of the intervention period.
Weight (in kilograms) Loss -- Post-intervention | 48-week period following the baseline period.
  Drop in weight from baseline to the end of the post-intervention period.
Change in Waist Measurement (in inches) -- Intervention | 36-week intervention period following the baseline period
  Change in waist measurements from baseline to the end of the intervention period.
Change in Waist Measurement (in inches) -- Post-intervention | 48-week period following the baseline period.
  Change in waist measurements from baseline to the end of the post-intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Teck H Ho, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Investigators will not be storing or sharing any personal identifiers. All individual level data will be anonymized, and only anonymized data will be shared with other researchers, upon request.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: After completion of all analysis. It will be made available in the supporting documentation.
Access Criteria: It will be made available in the supporting documentation.